CLINICAL TRIAL: NCT00438477
Title: A Preliminary Study To Explore Subareolar Injection As The Site For Lymphatic Mapping And Sentinel Lymph Node Biopsy In Patients With Breast Cancer
Brief Title: Injection Methods in Finding the Sentinel Lymph Node During Lymphatic Mapping and Sentinel Lymph Node Biopsy in Patients With Invasive Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ID01-538; P30CA016672 (NIH); MDA-ID-01538 (Other: UT MD Anderson Cancer Center); CDR0000355838 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — iso-sulfan blue; Technetium Tc 99m Sulfur Colloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Injection Methods (Experimental): One injection site with radioactive tracer intraparenchymal/peritumoral (around the tumor), and other subareolar (around the nipple)
  Interventions: Drug: Isosulfan Blue; Procedure: Lymphangiography; Radiation: Technetium Tc 99m sulfur colloid

INTERVENTIONS:
Drug: Isosulfan Blue — At time of surgery, breast injected with 3-5 cc of isosulfan blue in subareolar or peritumoral position.
  Other Names: lymphazurin
Procedure: Lymphangiography — 2 lymphoscintigraphy images performed following peritumoral and subareolar injection of breast
Radiation: Technetium Tc 99m sulfur colloid — At least 2 days before scheduled surgery, receive technetium Tc 99m sulfur colloid by peritumoral injection; and again the day before surgery by subareolar injection.
  At the time of surgery, patients receive isosulfan blue by subareolar injection.

SUMMARY:
RATIONALE: Diagnostic procedures, such as lymphoscintigraphy using an injection under the nipple or near the tumor, may help doctors find out how far the disease has spread.

PURPOSE: This clinical trial is studying two different injection methods to compare how well they find the sentinel lymph node during lymphatic mapping and sentinel lymph node biopsy in patients with invasive breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare subareolar injection with peritumoral injection in identifying the sentinel node during breast lymphatic mapping in patients with invasive breast cancer.
* Compare the lymphatic drainage patterns using lymphoscintigraphy of the breast with subareolar injection vs peritumoral injection.

OUTLINE: At least 2 days before scheduled surgery, patients receive technetium Tc 99m sulfur colloid by peritumoral injection followed by lymphoscintigraphy. Images are obtained at 30 minutes and after 2 and 3 hours, provided no drainage is noted. Patients then receive technetium Tc 99m sulfur colloid by subareolar injection followed by another lymphoscintigraphy.

At the time of surgery, patients receive isosulfan blue by subareolar injection. A handheld gamma probe is used to locate the sentinel node. If the sentinel node is identified, it is excised and the scheduled breast surgery is performed. If the sentinel node cannot be identified, patients undergo the scheduled breast surgery.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study within 12.5 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have either pathologic, radiologic or clinical evidence of breast cancer with invasion, suspicious for invasion or microinvasion.
2. Patients who are candidates for a total mastectomy or segmental mastectomy or axillary dissection.
3. Patients who have undergone neoadjuvant chemotherapy who have an FNA confirmed lymph node positive for metastatic disease prior to induction chemotherapy and are then found to have grossly palpable disease but are ultrasound node negative at time of study entry.
4. Patients must sign an informed consent and be registered before the procedure is performed.

Exclusion Criteria:

1. A pregnancy test will be required preoperatively in women of childbearing potential and patients who are pregnant will be excluded from this study.
2. Patients who have undergone neoadjuvant chemotherapy who have an FNA confirmed lymph node metastatic disease prior to induction chemotherapy and are then found to have grossly suspicious palpable disease and are ultrasound node positive at the time of study entry.
3. Patients with known allergy to isosulfan blue dye or any related compounds.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2005-06; Primary Completion 2006-08 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Lymphatic drainage patterns as determined by peritumoral and subareolar injections | 12 months to collect data
  Evaluate outcome descriptively.
Identification rate of sentinel nodes and negative predictive value associated with subareolar injection | 12 months to collecte data
  Evaluate outcome descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Gildy V. Babiera, MD, Study Chair — M.D. Anderson Cancer Center; Ebrahim Delpassand, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- M. D. Anderson Cancer Center at University of Texas, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org